CLINICAL TRIAL: NCT02914756
Title: Cognitive Impairment After Critical Illness, Links Between Sepsis, Cognitive Function and Non-resolving Inflammation
Brief Title: HMGB1 in ICU-survivors
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Peter Sackey, MD, PhD, Karolinska University Hospital
Other Study IDs: EPN 2013/1221-31/1
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Sepsis; Cognitive Impairment
MeSH Terms: conditions — Sepsis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis: Patients suffering from Severe sepsis or Septic chock at the ICU.
- Non-Sepsis: Patients being treated at ICU but not suffering from severe sepsis/septic chock

SUMMARY:
Is HMGB1 (High Mobility Group Box 1) elevated in sepsis patients for weeks after recovery from severe sepsis/septic shock, similar to what has been observed in mice? Do patients recovering from severe sepsis/septic shock suffer from cognitive impairment and is such impairment associated with prolonged HMGB1 levels in plasma? Is there a difference from patients recovering from critical illness without prior sepsis?

ELIGIBILITY:
Inclusion Criteria:

* Male/Female age 18-17
* Expected ICU-stay more than 24 hours

Exclusion Criteria:

* Dont understand the language
* Substance abuse, alcohol or drugs
* Blind, deaf or suffering from aphasia
* Ongoing psychiatric illness or psychopharmacological treatment
* Suffering from dementia och mentally impaired
* Structured brain damage or meningitis
* Palliative Care
* ICU-treated for more than 48 hours
* Transferred from other ICU
* Being treated with ECMO
* Not having residency in Stockholm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated at Karolinska University Hospital Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Is HMGB1 elevated in sepsis patients for weeks after recovery from severe sepsis/septic shock, similar to what has been observed in mice? | 2 years
Do patients recovering from severe sepsis/septic shock suffer from cognitive impairment and is such impairment associated with prolonged HMGB1 levels in plasma? Is there a difference from patients recovering from critical illness without prior sepsis? | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Surgical Services and Intensive Care Medicine, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Bruck E, Svensson-Raskh A, Larsson JW, Caravaca AS, Gallina AL, Eberhardson M, Sackey PV, Olofsson PS. Plasma HMGB1 levels and physical performance in ICU survivors. Acta Anaesthesiol Scand. 2021 Aug;65(7):921-927. doi: 10.1111/aas.13815. Epub 2021 Mar 27. PMID 33725363